CLINICAL TRIAL: NCT00821795
Title: Veterans Inpatient Insulin Study and Transition Algorithm: Efficacy of Insulin Analogs for Inpatient Glycemic Control and Transition to Outpatient Therapy
Brief Title: Veterans Inpatient Insulin Study and Transition to Outpatient Therapy
Acronym: VIISTA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dennis G. Karounos, M.D. (U.S. Federal Agency)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor-Investigator, Dennis G. Karounos, M.D., Chief, Endocrinology Section, Staff Physician, Lexington VA Medical Center
Organization: Lexington VA Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIISTA-596-1
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Results first posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus, Type 2; insulin; therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NPH/Regular 70/30 mix (Active Comparator): transition insulin therapy with NPH/Regular 70/30 mix for outpatient glycemic control following a hospitalization for non-critical acute illness
  Interventions: Drug: NPH/Regular 70/30 mix
- Aspart insulin analog biphasic mix (Active Comparator): transition insulin therapy with Aspart insulin analog 70/30 mix for outpatient glycemic control following a hospitalization for non-critical acute illness
  Interventions: Drug: insulin aspart protamine/insulin aspart 70/30 mix

INTERVENTIONS:
Drug: NPH/Regular 70/30 mix — injectable solution, subcutaneous,0.3-0.5 units/kg/day divided into twice per day dosage, 16 weeks duration
  Other Names: Novolin 70/30
  Arms: NPH/Regular 70/30 mix
Drug: insulin aspart protamine/insulin aspart 70/30 mix — injectable solution, subcutaneous, 0.3-0.5 units/kg/day divided into twice per day dosage, for 16 weeks
  Other Names: Novolog Mix 70/30
  Arms: Aspart insulin analog biphasic mix

SUMMARY:
Volunteers are being invited to take part in a research study about insulin therapy of diabetes. They are being invited to take part in this research study because they have diabetes and have an illness requiring hospitalization. If they volunteer to take part in this study, they will be one of about 120 people to do so. The investigators hope to answer the following research questions:

* To show that insulin aspart protamine 70/30 mix taken twice daily is as good as insulin NPH/Reg 70/30 mix taken twice a day for treatment of diabetes after discharge from the hospital.
* To show how safe the two medicines are (insulin aspart 70/30 mix vs. insulin NPH/Reg 70/30 mix) and how well they work for the treatment of diabetes when transitioning from inpatient therapy to outpatient care.

DETAILED DESCRIPTION:
By doing this study, we hope to learn the optimal way to use insulin therapy to treat individuals during a hospitalization for an illness as well as during the recovery phase of the illness for twenty-four weeks after discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes for duration of three-months or longer
* greater than or equal to 40 years of age
* Written informed consent to participate in the study
* Admitted for hospitalization at VA Medical Center Lexington, KY
* Able and willing to do the following:
* Use the insulin injection device provided to you as you are instructed
* Check your blood sugar as instructed using the blood sugar monitor and send the results by a glucose log or a telephone transmitter provided to you for use during the study
* Enter your information in a diary provided to you
* You have an acute non-critical medical illness requiring inpatient hospitalization (at least 24 hour admission) with a blood glucose between 140 and 400 mg/dl.
* You require further hospitalization after being released from intensive care unit for an acute illness

Exclusion Criteria:

* Have developed a severe illness requiring treatment in an intensive care unit as determined by your admitting physician.
* Are pregnant or intend to become pregnant during this study, or are a sexually active woman who could become pregnant and are not practicing a birth control method considered acceptable by your study doctor for preventing pregnancy.
* Are a woman who is breastfeeding.
* Have a history of heart disease that limits your physical activity
* Have had a kidney transplant or are currently receiving kidney dialysis
* Have history of cancer other than minor skin cancer.
* Have had a blood transfusion or severe loss of blood in the past 3 months or have any disease of the blood system.
* Are allergic or sensitive to study insulin.
* Are currently receiving oral steroid therapy.
* Are currently on any other investigational medications or investigational protocols
* Have drug or alcohol abuse that in the investigator's opinion would cause the individual to be non-compliant.
* Are poorly compliant with the currently prescribed diabetes regimen or self monitoring of blood glucose, as defined by the investigator.
* Have a mental condition that renders you unable to understand the scope and possible consequences of the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-03-11 (Actual); Primary Completion 2013-04-23 (Actual); Study Completion 2013-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis G Karounos, MD, Principal Investigator — VA Medical Center Lexington, KY and University of Kentucky College of Medicine
Locations (1):
- VA Medical Center - Lexington 596, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NPH/Regular 70/30 Mix | Aspart Insulin Analog Biphasic Mix
Started | 50 | 64
Completed | 44 | 60
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NPH/Regular 70/30 Mix | Aspart Insulin Analog Biphasic Mix | Total
Number analyzed (Participants) | 50 | 64 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (9) | 62.8 (8.6) | 63.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 50 | 62 | 112

OUTCOME MEASURES:

1. Primary Outcome: For Transition From Inpatient to Outpatient Care, Evaluate Glycemic Control in Subjects Randomized to Receive 70/30 NPH/Regular Insulin or Aspart Analog 70/30 Mix Bid- Main Outcome Will be HbA1c During Transition Outpatient Therapy Phase.
Description: Hemoglobin A1c
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: % hemoglobin A1c
Arm/Group | NPH/Regular 70/30 Mix | Aspart Insulin Analog Biphasic Mix
Number analyzed (Participants) | 44 | 60
% hemoglobin A1c | 8.32 (1.5) | 8.35 (1.95)

2. Secondary Outcome: Seven Point Blood Glucose Profiles
Description: mg/dl
Time Frame: 2 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Patient-reported Outcomes - Diabetes Symptom Checklist to Evaluate Perception of Diabetes Control
Time Frame: 16 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Hypoglycemia
Time Frame: daily
Reporting Status: Not Posted

5. Secondary Outcome: Twice Daily Blood Glucose Monitoring Using Telehealth Transmitter
Time Frame: daily
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | NPH/Regular 70/30 Mix | Aspart Insulin Analog Biphasic Mix
Serious Adverse Events (participants affected / at risk) | 15/50 | 10/64
Other Adverse Events (participants affected / at risk) | 6/50 | 9/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NPH/Regular 70/30 Mix (N=50) | Aspart Insulin Analog Biphasic Mix (N=64)
Cardiovascular disease (Cardiac disorders) | 7 (7) | 6 (6)
Cerebral vascular disease (Vascular disorders) | 1 (1) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Genitourinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Neurological disease (Nervous system disorders) | 1 (1) | 1 (1)
Pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Adverse reaction (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NPH/Regular 70/30 Mix (N=50) | Aspart Insulin Analog Biphasic Mix (N=64)
Severe Hypoglycemia (Metabolism and nutrition disorders) | 6 (6) | 9 (9)

LIMITATIONS AND CAVEATS:
The study is confined to Veterans requiring hospital admission for an acute medical illness on a general medicine ward with our study population being predominately elderly males greater than sixty years of age.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No